CLINICAL TRIAL: NCT01508702
Title: A Phase 3 Randomized, Double-Blind, Multicenter, Placebo- Controlled Study to Assess the Efficacy and Safety of Lesinurad Monotherapy Compared to Placebo in Subjects With Gout and an Intolerance or Contraindication to a Xanthine Oxidase Inhibitor
Brief Title: Lesinurad Monotherapy in Gout Subjects Intolerant to Xanthine Oxidase Inhibitors
Acronym: LIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDEA594-303; 2011-003756-39 (EudraCT Number)
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2015-07

CONDITIONS: Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lesinurad 400 mg (Experimental)
  Interventions: Drug: lesinurad
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lesinurad — Tablets, 400 mg QD
  Arms: lesinurad 400 mg
Drug: Placebo — Tablets, Placebo QD
  Arms: placebo

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of lesinurad compared to placebo in patients who are intolerant or have a contraindication to allopurinol or febuxostat.

DETAILED DESCRIPTION:
Allopurinol is the standard of care for the treatment of gout. In practice, approximately 20% of patients report side effects with allopurinol and 5% discontinue allopurinol due to side effects. Allopurinol can cause gastrointestinal intolerance, such as nausea and diarrhea, which appears to be dosedependent. Rash develops in about 2% of patients treated with allopurinol, and in about 20% of patients treated with allopurinol and ampicillin or amoxicillin. Allopurinol hypersensitivity syndrome remains a major concern among physicians. Mortality has been estimated to be up to nearly one quarter of AHS cases, with multiorgan system disease including hepatocellular changes and renal failure being a serious concern. Allopurinol is also relatively contraindicated for use in combination with 6-mercaptopurine and azathioprine, for which 1/4 to 1/3 lower doses must be given in order to avoid hematologic toxicity. Febuxostat, in clinical trials, has shown a similar AE profile to allopurinol. Liver function abnormalities, nausea, arthralgia and rash were the most commonly reported AEs. In postmarketing experience, Stevens Johnson Syndrome and hypersensitivity rashes have been reported (febuxostat prescribing information). Withdrawals due to AEs were similar in frequency to allopurinol as well. Relative contraindications in combination with 6-mercaptopurine and azathioprine are similar to allopurinol as well. Lesinurad may be an important therapeutic option for patients who either cannot tolerate or who have a contraindication to the use of allopurinol or febuxostat.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures, the risks involved and willing to provide written informed consent before the first study related activity.
* Subject meets the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has an sUA level ≥ 6.5 mg/dL at the Screening and Day -7 Visits.
* Subject must be able to take gout flare prophylaxis with colchicine or NSAID (including Cox-2 selective NSAID) ± PPI.
* Subject has a history (either by medical record or subject interview) of intolerance or a contraindication to either allopurinol or febuxostat.
* Body mass index (BMI) < 45 kg/m2

Exclusion Criteria:

* Subject who is taking any other approved urate-lowering medication that is indicated for the treatment of gout at the Screening Visit.
* Subject with a documented history or suspicion of kidney stones.
* Subject who is pregnant or breastfeeding.
* Subject who consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
* Subject with a history or suspicion of drug abuse within the past 5 years.
* Subject that requires or may require systemic immunosuppressive or immunomodulatory treatment.
* Subject with a known or suspected human immunodeficiency virus (HIV) infection.
* Subject with a positive test for active hepatitis B or hepatitis C infection.
* Subject with a history of malignancy within the previous 5 years with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia or treated in situ Grade 1 cervical cancer.
* Subject within the last 12 months with: unstable angina, New York Heart Association class III or IV heart failure, myocardial infarction, stroke, or deep venous thrombosis; or subjects currently receiving anticoagulants.
* Subject with uncontrolled hypertension.
* Subject with an estimated creatinine clearance < 30 mL/min.
* Subject with active peptic ulcer disease requiring treatment.
* Subject with active liver disease, or hepatic dysfunction.
* Subject receiving chronic treatment with more than 325 mg salicylates per day.
* Subject taking valpromide, progabide, or valproic acid.
* Subject who has received an investigational therapy within 8 weeks or 5 half-lives (whichever is longer) prior to the Screening Visit.
* Subject with any other medical or psychological condition, which in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Storgard, MD, Study Director — Ardea Biosciences, Inc.
Locations (100):
- United States (74):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Covina, California
  - Huntington Park, California
  - Irvine, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Englewood, Colorado
  - Milford, Connecticut
  - Trumbull, Connecticut
  - Boynton Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Plant City, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Newnan, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Chicago, Illinois
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - South Traverse, Michigan
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Southfield, Missouri
  - Washington, Missouri
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Hartsdale, New York
  - New Windsor, New York
  - New York, New York
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Willoughby Hills, Ohio
  - Norman, Oklahoma
  - Jenkintown, Pennsylvania
  - Lancaster, Pennsylvania
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Sellersville, Pennsylvania
  - Myrtle Beach, South Carolina
  - Rock Hill, South Carolina
  - Spartanburg, South Carolina
  - Brentwood, Tennessee
  - Spring Hill, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Victoria, Texas
  - South Bountiful, Utah
  - West Jordon, Utah
  - West Layton, Utah
  - Chesapeake, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
- Australia (3):
  - Butterfield, Queensland
  - Hobart, Tasmania
  - Tasmania
- Belgium (5):
  - Anderlecht, Brussels Capital
  - Genk, Limburg
  - Gozée
  - Kortrijk
  - Yvoir
- Canada (8):
  - Coquitiam, British Columbia
  - Coquitlam, British Columbia
  - Victoria, British Columbia
  - London, Ontario
  - Mississauga, Ontario
  - Toronto, Ontario
  - Québec, Quebec
  - Rimouski, Quebec
- Germany (3):
  - Dresden, Saxony
  - Leipzig, Saxony
  - Dresden
- New Zealand (2):
  - Tauranga, Bay of Plenty
  - Auckland
- South Africa (5):
  - Durban
  - Pretoria
  - Rondebosch
  - Stellenbosch
  - Thabazimbi

REFERENCES:
- [Derived] Topless R, Noorbaloochi S, Merriman TR, Singh JA. Change in serum urate level with urate-lowering therapy initiation associates in the immediate term with patient-reported outcomes in people with gout. Semin Arthritis Rheum. 2022 Oct;56:152057. doi: 10.1016/j.semarthrit.2022.152057. Epub 2022 Jun 29. PMID 35835008
- [Derived] Tausche AK, Alten R, Dalbeth N, Kopicko J, Fung M, Adler S, Bhakta N, Storgard C, Baumgartner S, Saag K. Lesinurad monotherapy in gout patients intolerant to a xanthine oxidase inhibitor: a 6 month phase 3 clinical trial and extension study. Rheumatology (Oxford). 2017 Dec 1;56(12):2170-2178. doi: 10.1093/rheumatology/kex350. PMID 29029210
- See also: Related Info — http://www.gouttrial.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lesinurad 400 mg: lesinurad 400 mg
Period: Overall Study
Arm/Group | Lesinurad 400 mg | Placebo
Started | 107 | 107
Completed | 84 | 94
Not Completed | 23 | 13
Not completed — Adverse Event | 7 | 3
Not completed — Gout flare | 2 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lesinurad 400 mg | Placebo | Total
Number analyzed (Participants) | 107 | 107 | 214
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (12.5) | 55.3 (12.0) | 54.4 (12.2)
Age, Customized [Number; unit: Participants]
  <65 | 87 | 80 | 167
  >=65 | 20 | 27 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 98 | 97 | 195
Region of Enrollment [Number; unit: Participants]
  Australia | 1 | 1 | 2
  Belgium | 5 | 4 | 9
  Canada | 5 | 6 | 11
  Germany | 5 | 2 | 7
  New Zealand | 3 | 2 | 5
  South Africa | 12 | 11 | 23
  United States | 76 | 81 | 157

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an sUA Level That is < 6.0 mg/dL
Time Frame: 6 months
Population: ITT Population
Measure: Number; unit: Number of Subjects
Units Other Than Participants: Subjects
Groups:
- Placebo: Placebo qd
Arm/Group | Lesinurad 400 mg | Placebo
Number analyzed (Participants) | 107 | 107
Number analyzed (Subjects) | 107 | 107
Number of Subjects | 32 | 2
Statistical Analysis 1: Comparison: Lesinurad 400 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.28, 95% CI 2-sided [0.19 to 0.37]

ADVERSE EVENTS:
Arm/Group | Lesinurad 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/107 | 4/107
Other Adverse Events (participants affected / at risk) | 39/107 | 8/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 400 mg (N=107) | Placebo (N=107)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lesinurad 400 mg (N=107) | Placebo (N=107)
Constipation (Gastrointestinal disorders) | 6 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 6 (6)
Oedema peripheral (General disorders) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 2 (2)
Blood creatinine increased (Investigations) | 9 (10) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 4 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.